CLINICAL TRIAL: NCT06263036
Title: Morphometric Examination of the Larynx
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Sevgi Bilgen, Associate Professor, Acibadem University
Other Study IDs: Bilgen S
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Laryngeal Dimensions in Males and Females
Keywords: larynx, measurement, cadaver, Turkish population
MeSH Terms: conditions — Laryngeal Diseases; Cadaver | interventions — Menogaril

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men: Cadavra
  Interventions: Other: Men; Other: Women
- Women: Cadavra
  Interventions: Other: Men; Other: Women

INTERVENTIONS:
Other: Men — Laryngeal cartilages
Other: Women — Laryngeal cartilages

SUMMARY:
Objective: To measure laryngeal dimensions in a sample of Turkish cadavers including males and females of various ages and heights.

Patients and Methods: Morphological measurement was performed on 102 laryngeal specimens. Laryngeal cartilages were collected from human cadavers. All dimensions of the cartilages were measured using a thread and vernier calipers. Age, sex, and height were recorded. Results for men and women were compared.

ELIGIBILITY:
Inclusion Criteria:human cadavers -

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Turkish cadavers including males and females of various ages and heights
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
To measure laryngeal dimensions in cadavers | 5 months
  To measure laryngeal dimensions in a sample of Turkish cadavers